CLINICAL TRIAL: NCT04111081
Title: Pilot Study of Clinical Randomized Controlled Trial of Auricular Pressure Therapy for Intervention of Postoperative Pain of Hemorrhoidectiomy
Brief Title: Auricular Pressure for Postoperative Pain After Hemorrhoidectiomy: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CXTD1701
Record Dates: First submitted 2019-09-17; First posted 2019-10-01 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Postoperative Pain
Keywords: hemorrhoidectiomy; postoperative pain; auricular pressure
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular pressure (Experimental): Use wangbuliuxing seed to stimulate auricular acupuncture point.
  Interventions: Other: Auricular pressure
- Sham auricular pressure (Sham Comparator): Use wangbuliuxing seed to stimulate auricular acupuncture point.
  Interventions: Other: Shame auricular pressure

INTERVENTIONS:
Other: Auricular pressure — Select related auricular points: Shenmen(TF4), sympathetic(AH6a), rectum(HX2), anus(HX5), stomach(CO4), subcortical(AT4). The auricle skin of the patient was disinfected 24 hours after the operation, and wanghuoxing seed will be used for stimulation. Ask patients press every two hours for one minute at each point. When the pain is severe, do pressure compressions at each point for 2 minutes once hour.
  Arms: Auricular pressure
Other: Shame auricular pressure — Select unrelated auricular points: eye(LO5), occipital(AT3), tonsil(LO7,8,9), lower auricular root(R3), dorsum auricular kidney(P5) and dorsum auricular lung(P2). The auricle skin of the patient was disinfected 24 hours after the operation, and wanghuoxing seed will be used for stimulation. Ask patients press every two hours for one minute at each point. When the pain is severe, do pressure compressions at each point for 2 minutes once hour.
  Arms: Sham auricular pressure

SUMMARY:
Auricular pressure is effective for postoperative analgesia after hemorrhoidectomy, but the evidence is not sufficient.

DETAILED DESCRIPTION:
This is a randomized, double-blind study to study the analgesic effect of auricular pressure pill on persistent pain after hemorrhoidectiomy. Baseline pain intensity scores (VAS>3) of the subjects will be collected 24 hours after the operation of the patients. Eligible subjects will be randomly assigned to receive auricular pressure pills or sham-auricular pressure pills. The treatment will last 5-7 days. Participants will receive auricular pressure once two days, and receive VAS, concomitant medication, PONV intensity scale and peripheral edema were recorded daily, and after the operation 24 hours, 3 days and 7 days the patients will receive anxiety and depression scale(HAD) , and VAS data will be collected by telephone at 3 and 6 months after the operation.

The statistical analysis results will be subject to the full analysis set (FAS) results, and a sensitivity analysis will be performed comparing the per-protocol (PP). The main indicators will be analyzed by covariance analysis, with VAS results as the dependent variable, grouping as the random factor, and age, course of disease, surgical method and baseline as the covariables to correct the P value. The secondary indicator analgesic usage rate will be analyzed using logistic regression analysis. Whether analgesic will be used as a dependent variable, grouping as a random factor, and age, course of disease, surgical method and evaluation time point will be analyzed as covariables. Other outcome indicators will be analyzed by covariance analysis, and the model will be the same as that of the main indicators. P<0.05 considered as significant difference, and SPSS20.0 used for analysis.

The purpose of this study was to seek high quality evidence-based medical evidence for intervention of auricular pressure pills on postoperative pain of hemorrhoidectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of grade II-IV mixed hemorrhoids and meet the operation conditions;
2. Age 18~65;
3. External stripping and internal ligation of mixed hemorrhoids, general anesthesia or lumbar shu point anesthesia;
4. VAS score ≥3 points after the implementation of analgesia pump;
5. Improve clinical auxiliary examination and sign informed consent.

Exclusion Criteria:

1. Combined with inflammatory hemorrhoids, thrombotic hemorrhoids, perianal eczema, perianal abscess and other perianal diseases that affect the evaluation of curative effect;
2. Combined with intestinal infectious diseases, intestinal polyps, rectal malignant tumors, etc;
3. Combined with severe cardiovascular disease, immune deficiency, mental disorder, or severe liver and kidney dysfunction;
4. Auricle skin lesions or auricle skin allergy to tape is difficult to tolerate treatment;
5. Combined cognitive impairment could not complete the efficacy; evaluation;
6. Pregnancy or planned pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale(VAS) | Day 1 after randomization.
  It is a unidimensional measure providing a simple solution for measuring subjective experience. The VAS scale is a 10-cm line with 0 cm indicating no symptoms and 10 cm indicates the greatest extent of symptoms. Twenty-four hours after the operation, VAS>3 in the case of an analgesic pump can be included in the randomized control group.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression scale(HAD) | Twenty-four hours, three days, and seven days after surgery
  The HAD scale included measures of anxiety and depression, with scores ranging from 0 to 21. 0-7 points means asymptomatic;A score of 8-10 means suspicious;A score of 11 to 21 means definitely symptomatic( anxiety or depression).
The utilization rate of analgesic drugs(Diclofenac Sodium Dual Release Enteric-coated Capsules) | Day 7 after randomization.
  The ratio of patients using analgesic drugs in each group was calculated (Patients who take bisphenolics once are considered users), and the utilization rate = number of users/total number of users ×100%.
Amount of analgesic drugs (Diclofenac Sodium Dual Release Enteric-coated Capsules) | Day 7 after randomization.
  The total analgesic drugs dose of each group was was considered as the amount of analgesics in the group.

OTHER OUTCOMES:
Tissue edema | Day 3, day4, day5, day6 and day7 after randomization.
  The degree of tissue edema was observed and recorded truthfully.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zheng, PhD, Principal Investigator — Chengdu University of Traditional Chinese Medicine
Locations (1):
- Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan, China